CLINICAL TRIAL: NCT02693340
Title: Evolution of Lymphocyte Populations Under Biotherapy in Inflammatory Bowel Disease
Acronym: IBDOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P150702
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — • Sampling period(s):
  * Blood: W0, W6, W14, W30 and W52 and relapse.
  * Biopsies and fecal: W0, W14 and M52 and relapse.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: sampling — • Sampling period(s):
  * Blood: W0, W6, W14, W30 and W52 and relapse.
  * Biopsies and fecal: W0, W14 and M52 and relapse.

SUMMARY:
This is a monocentric prospective study for the collection of biological samples (blood and biopsies) to be used for in vitro biomarker assay(s) performed to identify predictive markers of response to biological treatments in inflammatory bowel disease (IBD).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more.
* Crohn's Disease Diagnosis (CD) or ulcerative colitis (UC) according to defined criteria (ECCO recommendations).
* Active disease as defined by clinical biological and/or morphological assessment.
* Initiation of an anti-Tumor Necrosis Factor (TNF) therapy (Infliximab, Adalimumab, Golimumab) or new biotherapy (Vedolizumab, Ustekinumab) provided in connection with the management of digestive disease.
* Patient (e) have signed and dated consent of the study before undertaking procedures related to the study.

Exclusion Criteria:

* Patients under guardianship / curators
* Following Situations

  * Persons unable to understand, read and / or sign an informed consent
  * Patient with the following functions: investigator or co-investigator, research assistant, pharmacist, study coordinator or having any involvement in the study
  * Uncooperative person or potentially non-compliant for the study and its procedures with predictable difficulties regular monitoring of over 1 year.
  * No affiliation to a social security scheme, a universal medical coverage or any similar plan.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's Disease Diagnosis (CD) or ulcerative colitis (UC)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Response to biological treatments | 12 months

SECONDARY OUTCOMES:
Microbiota variation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Allez, MD PhD, Principal Investigator — APHP
Locations (1):
- Gastroenterology department, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Veyssiere M, Hammoudi N, Le Bourhis L, Hassid D, Bonnet J, Tran Minh ML, Baudry C, Gornet JM, Chardiny V, Seksik P, Nancey S, Carbonnel F, Treton X, Wils P, Buisson A, Boureille A, Hebuterne X, Serrero M, Fumery M, Louis E, Blanc P, Peyrin-Biroulet L, Bezault M, Soumelis V, Allez M. Blood proteomic signatures associated with disease activity in inflammatory bowel diseases. J Crohns Colitis. 2025 Sep 28;19(9):jjaf162. doi: 10.1093/ecco-jcc/jjaf162. PMID 40920365